CLINICAL TRIAL: NCT06731712
Title: Targeted Physical Function Exercises on Frailty and Falls Management in Pre-Frail Community-Dwelling Older Adults: a Randomized Controlled Trial
Brief Title: Targeted Physical Function Exercises on Frailty and Falls Management in Pre-Frail Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Mediterranean University (Other)
Responsible Party: Principal Investigator, Konstantinos Giakoumidakis, Associate Professor, Hellenic Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3589/2020
Record Dates: First submitted 2024-10-26; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Frailty Syndrome; Pre-frail Older Adults
Keywords: Frailty; Concerns about Falling; Physical Function exercises
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Function Group (Experimental): Physical function interventions including strength, balance, and mobility exercises
  Interventions: Other: Physical Function Exercises
- Control Group (No Intervention): Will continue their normal lives

INTERVENTIONS:
Other: Physical Function Exercises — Physical function interventions included strength, balance, and mobility exercises. More specifically, the exercises include progressively increasing intensity strengthening exercises with a resistance band for the following muscle groups: hip abductor and extensor muscles, knee flexor and extensor muscles, and shoulder abductor and external rotator muscles. Other exercises consist of standing calf raises, squats, bridges, and push-ups. Additionally, functional exercises include heel-to-toe standing or walking, single-leg standing, stepping over obstacles, bending down, and lifting an object with feet together.
  Other Names: Targeted Physical Function Exercises
  Arms: Physical Function Group

SUMMARY:
The investigators will conduct a randomized controlled trial to assess the impact of targeted physical function exercises on frailty and falls in community-dwelling adults over 65 years of age. Participants will be randomized to an intervention and a control group to undergo an 18-month assessment.

The hypothesis of this study is to investigate the impact of targeted physical function exercises on managing frailty status and concerns about falling among pre-frail older adults. By implementing individualized intervention programs tailored to improve strength, balance, and mobility, the investigators aim to enhance physical function and reduce the risk of frailty-related adverse health outcomes. The investigators seek to empower pre-frail older adults to proactively manage their health, maintain independence, and improve their quality of life as they age.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 65 and over
* classified as pre-frail according to SHARE-Frailty Instrument
* independent of movement and activity
* able to perform Mini-Mental Status Examination (MMSE) score ≥24

Exclusion Criteria:

* severe contraindications for physical exercise
* central nervous system impairments
* inability to speak and understand Greek properly
* a cognitive state that prevents understanding the researcher's instructions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Level of Frailty status | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  SHARE Frailty Instrument will be used. Diagnostic criteria include involuntary loss of weight and muscle mass, exhaustion, low physical activity, slowness, and reduced grip strength. The presence of three or more criteria indicates frailty, while the presence of less than three pre-frailty
Concerns about Falling | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  The Falls Efficacy Scale - International (FES-I), a 16-item questionnaire that assesses the participant's fall efficacy, will be used to measure the level of concern about falling during various social and physical activities. Every item has a four-point (1-4) score, summarizing a total score of 64 points. A 16-22 score indicates low concern about falling, and a 23-64 high concern.

SECONDARY OUTCOMES:
Physical Performance | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  The Short Physical Performance Battery (SPPB) will be used to assess physical performance. It is an assessment tool consisting of 3 tests in three different domains (walking, sit-to-stand, and balance) to assess function: a 3- or 4-meter walking time at the usual speed, one single chair stand, and time to complete five chair stands, and three balance tests of progressive difficulty, holding for 10 seconds (side-by-side, semi-tandem, tandem stand). Each test is rated on a scale of 0 to 4, summed to give an overall score ranging from 0 to 12, with a higher score indicating better performance.
Functional Mobility | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  For quantifying functional mobility, the Time Up and Go test (TUG) will be used. Participants will be observed and timed while standing up from an armchair, walking three meters, making a turn, and returning to their sitting position. The timer will start when the participants are ready to stand up and stop when they return sitter.
Functional Balance | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  The Berg Balance Scale (BBS) will be used to assess a participant's ability to balance safely during specific tasks. It evaluates dynamic and static balance through 14 functional tasks, with each task answered on a five-point scale ranging from 0, indicating the lowest level of functioning, to 4, the highest level of functioning. The final summary score ranges from 0 to 56.
Quality of Daily Living | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  To assess the quality of life of the participants, the WHOQOL-BREF scale will be used, which includes 26 items concerning 4 domains of health (physical health, psychological health, social relationships, and environment) and 4 additional items concerning nutrition, satisfaction with work, home life, and social life. Each item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100 scale.
Depression | From baseline (T0), at 6 months (T1), at 12 months (T2), to the end of the intervention at 18 months (T3).
  The short-form Geriatric Depression Scale (GDS), consisting of 15 yes-or-no questions with a total score range of 0 to 15, was used to assess the participant's depressive symptoms. A score of 0 to 5 is normal. A score greater than 5 suggests depression.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Giakoumidakis, Principal Investigator — Hellenic Mediterranean University
Locations (1):
- Hellenic Mediterranean University, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No